CLINICAL TRIAL: NCT00626184
Title: A Phase 1, Two Stage, Single Dose, Single-Blind, Placebo Controlled, Dose Escalation, Crossover Study of the Safety and Tolerability of ALV003 in Healthy Adult Volunteers and Subjects With Well-Controlled Celiac Disease
Brief Title: A Phase 1, Study of the Safety and Tolerability of ALV003 in Healthy Adult Volunteers and Subjects With Well-Controlled Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Vijaya Pratha, M.D., Principal Investigator, Clinical Applications Laboratories Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ALV003-0811
Record Dates: First submitted 2008-02-13; First posted 2008-02-29 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Celiac Disease
Keywords: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Placebo
  Interventions: Drug: 4 dose levels of ALV003
- B (Active Comparator): Active study Drug: ALV003
  Interventions: Drug: 4 dose levels of ALV003

INTERVENTIONS:
Drug: 4 dose levels of ALV003 — 4 dose levels of ALV003 vs placebo
  Other Names: ALV003 and ALV003 placebo equivalent

SUMMARY:
To assess safety and tolerability of ALV003 in healthy volunteers and patients with Celiac Disease

DETAILED DESCRIPTION:
A Phase 1, Two Stage, Single Dose, Single-Blind, Placebo Controlled, Dose Escalation, Crossover Study of the Safety and Tolerability of ALV003 in Healthy Adult Volunteers and Subjects With Well-Controlled Celiac Disease

ELIGIBILITY:
INCLUSION

* Health Status

  1. Healthy volunteers must be in good health
  2. Celiac Disease must be well controlled and in good health
* Either male or non-lactating, non-pregnant females who are postmenopausal, sterile or using at least two acceptable and highly effective birth control methods.
* Body Mass Index (BMI) of < 30 kg/m2,

EXCLUSION

* A positive urine test for alcohol or illegal drugs at screening.
* The subject has received an experimental drug within 30 days of the present study.
* History of substance abuse, within the last 5 years
* Clinically significant abnormal lab values, as determined by the PI
* Alcohol consumption of > 2 standard drinks equivalents per day12. Positive pregnancy test within 7 days prior to study drug administration.
* history of any medically significant condition considered by the PI to adversely affect participation in the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | Throughout

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Pratha, MD, Principal Investigator — Clinical Applications Laboratory Inc.
Locations (1):
- Clinical Applications Laboratories Inc., San Diego, California, United States